CLINICAL TRIAL: NCT06528613
Title: Real World Study in Greek Patients with BPH for the Evaluation of Disease Control and QoL Under FDC Treatment with Solifenacin/tamsulosin
Brief Title: Real World Study in Greek Patients with BPH for Disease Control and QoL Under FDC Treatment with Solifenacin/Tamsulosin.
Acronym: KALLIRROI
Status: Recruiting | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Elpen Pharmaceutical Co. Inc.
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Benign prostatic hyperplasia (BPH) is an age-related progressive condition of the prostate gland that results in an increase in prostate size.

Although the "normal" prostate in adult men usually has a volume of 15-30 ml, a value above 30 ml is usually considered "enlarged". However, the threshold at which a prostate is considered enlarged has not been strictly defined and therefore for many physicians an enlarged prostate is a subjective finding on examination.

BPH can only be defined histologically (increase in the number of epithelial cells and stromal cells), but in clinical practice it is characterized by lower urinary tract symptoms [LUTS]. The disease leads to increased pressure in the urethra, causing resistance to urine flow, known as Bladder Outlet Obstruction (BOO). This resistance can also lead to changes in bladder function caused by the obstruction, such as overactivity of the bladder detrusor muscle or, conversely, reduced detrusor contractility. BOO can present as LUTS, infections or retention, as well as other conditions.

LUTS can be divided into storage (irritant), obstructive (urinary) and post-urinary symptoms and appear frequently causing intense discomfort, reducing the quality of life. LUTS are traditionally associated with bladder outlet resistance (BOO), most commonly when histologic BPH progresses through benign prostatic enlargement (BPE) to benign prostatic obstruction (BPO).The European Urological Association (EAU) reports that LUTS are a common problem in adult men with a significant impact on quality of life (QoL). Accordingly, he suggests the use of the a1-blocker/muscarinic receptor antagonist combination in men with moderate to severe storage symptoms, voiding symptoms and PVR < 150 ml, in order to reduce the risk of acute urinary retention and relieve irritants. (storage) symptoms, leading to an improvement in the patient's quality of life. Given the small abundance of data for patients in Greece with BPH, this study will evaluate the fixed combination of solifenacin/tamsulosin in terms of disease control and improvement of the quality of life of patients with BPH. Before enrolling in the study and before signing the consent form, patients must have already received the drug with solifenacin/tamsulosin and then they are enrolled in the observational study where the physician applies his/her standard clinical practice.

DETAILED DESCRIPTION:
The only clearly defined risk factors for BPH are age and the presence of elevated androgens in the blood. But there are other factors that can influence the prevalence of clinical disease such as metabolic syndrome, diabetes, obesity, hypertension, diet and heredity.

Clinical BPH often occurs within the same family. If one or more first-degree relatives have had BPH, then a person is at greater risk of developing the disease. The probability of developing BPH and the rates of occurrence and progression of LUTS increase significantly with age. In a study of 278 men with an average age of 58 years, it was shown that prostate volume increased at an average rate of 0.6ml per year.

Although the severity of symptoms cannot be directly related to prostate volume, having a large prostate volume is a risk factor for developing LUTS (a larger prostate is associated with an increased risk of urinary retention).

Data support that the metabolic syndrome may influence the natural course regarding the development of BPH and BOO. Metabolic syndrome includes hypertension, dyslipidemia, glucose intolerance, obesity, and insulin resistance with compensatory hyperinsulinemia.

In a meta-analysis it was shown that the obese, the elderly, patients with low HDL cholesterol values and patients with metabolic syndrome had a significantly higher total prostate volume.

Diabetes mellitus as a cause of bladder dysfunction can manifest either as overactivity or as poor detrusor function. Diet has been reported as a risk factor for the development of BPH. High amounts of vegetables and soy products in the diet may explain the lower rate of BPH in Eastern compared to Western countries. The association of alcohol, diet, and other lifestyle factors with obstructive uropathy was investigated in a cohort of 6,581 Japanese-American men, 846 of whom were later diagnosed with BPH (after 17 years of follow-up). Total alcohol intake was inversely associated with the risk of developing obstructive uropathy or BPH (i.e., reduced risk of developing the disease).

In the present study purpose is to evaluate the symptoms of the lower urinary tract in patients with BPH; the International Prostate Symptom Score (IPSS) questionnaire will be used, which is a modification of the AUA Symptom Index by adding a question that evaluates the quality of life in relation to the disease.

Both the AUA index and the IPSS questionnaire, although not specific for BPH, prostate volume, urine flow rate, residual urine volume after voiding or bladder obstruction, have been validated and are sufficiently sensitive for be used in symptom assessment and treatment selection. Although the assessment of specific symptoms is necessary for the treatment outcome of LUTS due to BPH, it is also important to have a simpler approach that addresses the patients' perception of the severity and change of their symptoms.

The Patient Global Impression of Severity (PGI-S) questionnaire assesses the patient's overall impression of the severity of his condition due to BPH symptoms and is a record of perception of the patient in a simple, valid and easily administered manner in clinical practice. The Patient Global Impression of Change (PGI-C) is the questionnaire it assesses the patient's overall impression of the change in their condition due to a treatment choice and is widely used in studies to assess chronic pain and/or for the patient's self-assessment of the overall improvement of a treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male adult patient with moderate to severe symptoms of BPH receiving monotherapy and not responding adequately.
* Male adult patient with BPH who has fully understood the study procedures and signed an informed consent form.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological male adult patient
Study Population: Male adult patients with moderate to severe symptoms of BPH received monotherapy and did not respond adequately and are receiving FDC of Solifenacin/Tamsulosin.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The assessment of disease control (BPH) and quality of life of patients. | 6 months
  The change in the total score (questions 1-7) and the quality-of-life question score of the International Prostate Symptom Score (IPSS) questionnaire after six months of treatment with a fixed combination of solifenacin/tamsulosin. The total disease control score is calculated by summing the scores of the seven symptom-related questions.
  In particular :
  Questions 1-6: 6-point response scale from 0 (not at all) to 5 (almost always). Question 7: 6-point response scale from 0 (none) to 5 (5 or more).
  This gives an overall score ranging from 0 to 35 where :
  0-7: mildly symptomatic, 8-19: moderately symptomatic, 20-35: severely symptomatic. Concerning the quality-of-life question score : 7-point response scale from 0 (no impact on QOL) to 6 (high impact on QOL).

SECONDARY OUTCOMES:
The assessment of patients' overall impression of their condition from Benign Prostatic Hyperplasia (BPH). | 6 months
  Assessment from baseline and after six months of solifenacin/tamsulosin fixed-combination treatment of the patient's global impression of change in severity and overall impression of change in condition due to BPH using the PGI- S (Patient Global Impression of Severity) and PGI-C (Patient Global Impression of Change), respectively.
  The Patient Global Impression of Change (PGI-C) scale measured patients' ratings of overall change in condition due to BPH compared to study baseline and range from 0 [very much better] to 7 [very much worse].
  The Patient Global Impression of Severity (PGI-S) scale measured patients' ratings of overall severity compared to study baseline and range from none to 7 very severe).
Assessment of the safety of the solifenacin/tamsulosin fixed dose combination during the study. | 6 months
  The recording of Adverse Events (AE) if they occur during the study. All directly observed adverse events and all adverse events (ΑΕ) spontaneously reported by the patient will be recorded, using accurate and comprehensive medical terminology. The ΑΕ reporting period for this study will begin at the 1st (selection) visit after the patient signs the informed consent form and end at the final follow-up visit. All AEs occurring during the adverse event reporting period must be reported, whether or not the event is considered to be related to the study drug. In all cases, the investigator should indicate whether there is a causal relationship between the reported event and the investigational medicinal product. In addition, any adverse event occurring after the adverse event reporting period that the investigator considers to be possibly related to the study drug should also be reported as an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Ginis, Study Director — Elpen Pharmaceutical Co. Inc.
Locations (6):
- Greece (6):
  - Second Department of Urology, Sismanoglio Hospital, Athens, Greece., Athens, Greece
  - Department of Urology, Venizelio General Ηospital, Heraklion, Greece
  - Department of Urology, General Hospital of Messinia, Kalamata, Greece
  - Department of Urology, General Hospital of Larissa, Larissa, Greece
  - Department of Urology, University Hospital of Rion, Pátrai, Greece
  - First Department of Urology, School of Medicine, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shibata K, Hirasawa A, Moriyama N, Kawabe K, Ogawa S, Tsujimoto G. Alpha 1a-adrenoceptor polymorphism: pharmacological characterization and association with benign prostatic hypertrophy. Br J Pharmacol. 1996 Jul;118(6):1403-8. doi: 10.1111/j.1476-5381.1996.tb15552.x. PMID 8832064
- [Background] Lepor H. Pathophysiology of benign prostatic hyperplasia in the aging male population. Rev Urol. 2005;7 Suppl 4(Suppl 4):S3-S12. PMID 16986052
- [Background] Ekman P. The prostate as an endocrine organ: androgens and estrogens. Prostate Suppl. 2000;10:14-8. No abstract available. PMID 11056488
- [Background] GBD 2019 Benign Prostatic Hyperplasia Collaborators. The global, regional, and national burden of benign prostatic hyperplasia in 204 countries and territories from 2000 to 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Healthy Longev. 2022 Nov;3(11):e754-e776. doi: 10.1016/S2666-7568(22)00213-6. Epub 2022 Oct 20. PMID 36273485
- [Background] Johnson TV, Abbasi A, Ehrlich SS, Kleris RS, Owen-Smith A, Raison CL, Master VA. IPSS quality of life question: a possible indicator of depression among patients with lower urinary tract symptoms. Can J Urol. 2012 Feb;19(1):6100-4. PMID 22316511
- [Background] Viktrup L, Hayes RP, Wang P, Shen W. Construct validation of patient global impression of severity (PGI-S) and improvement (PGI-I) questionnaires in the treatment of men with lower urinary tract symptoms secondary to benign prostatic hyperplasia. BMC Urol. 2012 Nov 7;12:30. doi: 10.1186/1471-2490-12-30. PMID 23134716